CLINICAL TRIAL: NCT04128319
Title: An Open-Label, Single-Arm, Multicenter Study, of Combination Anti-CD3/CD7 Immunotoxin (T-Guard) for Steroid-Refractory Acute Graft-versus-Host Disease)
Brief Title: T-Guard as Treatment for Steroid Refractory Acute GVHD (BMT CTN 1802)
Acronym: 1802
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Initiated a new randomized trial per discussion with FDA
Sponsor: Xenikos (Industry)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Cancer Institute (NCI) (NIH); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN1802; 2U10HL069294-11 (NIH); 5U24HL138660 (NIH)
Record Dates: First submitted 2019-09-27; First posted 2019-10-16 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Steroid-Refractory Acute Graft Versus Host Disease
Keywords: Steroid-refractory acute GVHD; Acute GVHD; GVHD treatment

STUDY DESIGN:
Intervention Model Description: A single group of patients will receive T-Guard for treatment of steroid-refractory acute GVHD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- T-Guard Treatment (Experimental): Patients will receive T-Guard for treatment of steroid-refractory acute GVHD.
  Interventions: Drug: T-Guard

INTERVENTIONS:
Drug: T-Guard — Patients will receive 4 doses of T-Guard treatment, administered intravenously as four 4-hour infusions at least two calendar days (no less than 40 hours) apart. Each dose consists of 4 mg/m^2 Body Surface Area (BSA).

SUMMARY:
The study is designed as an open-label, single arm Phase III, multicenter trial to evaluate the efficacy and safety of T-Guard treatment in patients with Steroid-Refractory acute Graft versus Host Disease (SR-aGVHD).

DETAILED DESCRIPTION:
Allogeneic Hematopoietic Cell Transplantation (allo-HSCT) is a potent immunotherapy with curative potential for several hematological disorders. Improvements in survival following allo-HSCT have led to its increasing use, but the leading cause of non-relapse mortality (NRM) remains graft-versus-host-disease (GVHD. Despite recent advances in the understanding of transplantation immune tolerance, aGVHD is a frequent and major complication of allo-HSCT involving activation of donor T-lymphocytes, which ultimately causes host tissue damage. T-Guard has a rapid onset, preferential killing of activated T cells, and short half-life, leading to depletion of allo-reactive T cells and quick post-treatment reconstitution of the immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 12.0 years of age at the time of consent.
2. Patient has undergone first allo-HSCT from any donor source using bone marrow, peripheral blood stem cells, or cord blood. Recipients of nonmyeloablative, reduced intensity, and myeloablative conditioning regimens are eligible.
3. Patients diagnosed with SR-aGVHD after allo-HSCT. SR is defined as aGVHD that:

   * Progressed after 3 days of primary treatment with prednisone (or equivalent) of greater than or equal to 2mg/kg/day
   * No improvement after 7 days of primary treatment with prednisone (or equivalent) of greater than or equal to 2mg/kg/day.
   * Patients with visceral (GI and/or liver) plus skin aGVHD at prednisone (or equivalent) initiation with improvement in skin GVHD without any improvement in visceral GVHD after 7 days of primary treatment with prednisone (or equivalent) of greater than or equal to 2mg/kg/day
   * Previously was treated with prednisone (or equivalent) of greater than or equal to 1mg/kg/day and aGVHD has developed in a previously uninvolved organ system

   Progression and no improvement are defined in the protocol. Improvement or progression in organs is determined by comparing current organ staging to staging at initiation of prednisone (or equivalent) treatment. Staging is performed per MAGIC criteria.
4. Evidence of myeloid engraftment (e.g., absolute neutrophil count greater than or equal to 0.5 × 10^9/L for 3 consecutive days if ablative therapy was previously used). Use of growth factor supplementation is allowed.
5. Patients or an impartial witness (in case the patient is capable of providing verbal consent but not capable of signing the informed consent form (ICF)) should have given written informed consent. For patients less than 18 years of age, a written informed consent of the parents or guardian and written assent of the patient will be obtained, per the local requirements.

Exclusion Criteria:

1. Patients who have been diagnosed with overlap syndrome, that is, with any concurrent features of cGVHD.
2. Patients requiring any of the following: mechanical ventilation, vasopressor support, or hemodialysis.
3. Patients who have received any systemic treatment, besides steroids, as upfront treatment of aGVHD OR as treatment for SR-aGVHD.
4. Patients who have severe hypoalbuminemia, with an albumin of less than or equal to 1 g/dl.
5. Patients who have a CK level of greater than 5 times the upper limit of normal.
6. Patients with uncontrolled infections. Infections are considered controlled if appropriate therapy has been instituted and, at the time of enrollment, no signs of progression are present. Progression of infection is defined as hemodynamic instability attributable to sepsis, new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
7. Patients with evidence of relapsed, progressing or persistent malignancy.
8. Patients with evidence of minimal residual disease requiring withdrawal of systemic immune suppression
9. Patients with known hypersensitivity to any of the components murine monoclonal antibodies (mAb) or Recombinant Ricin Toxin A-chain (RTA).
10. Patients who have received more than one allo-HSCT.
11. Patients with known human immunodeficiency virus infection.
12. Female patients who are pregnant, breast feeding, or, if sexually active and of childbearing potential, unwilling to use effective birth control from start of treatment until 30 days after the last infusion of T-Guard.
13. Male patients who are, if sexually active and with a female partner of childbearing potential, unwilling to use effective birth control from start of treatment until 65 days after the last infusion of T-Guard.
14. Patients with any condition that would, in the investigator's judgment, interfere with full participation in the study, including administration of study drug and attending required study visits; pose a significant risk to the patient; or interfere with interpretation of study data.
15. Patients whose decision to participate might be unduly influenced by perceived expectation of gain or harm by participation, such as patients in detention due to official or legal order.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehdi Hamadani, MD, Principal Investigator — Medical College of Wisconsin; John Levine, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Gabrielle Meyers, MD, Study Chair — Oregon Health and Science University
Locations (24):
- United States (24):
  - City of Hope National Medical Center, Duarte, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Indiana University, Indianapolis, Indiana
  - University of Kansas, Westwood, Kansas
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Mount Sinai Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Meyers G, Hamadani M, Martens M, Ali H, Choe H, Dawson P, Harris AC, van Hooren E, Klaassen W, Leifer E, MacMillan ML, van Oosterhout Y, Perez L, Pusic I, Vo P, Levine JE. Lessons learned from early closure of a clinical trial for steroid-refractory acute GVHD. Bone Marrow Transplant. 2022 Feb;57(2):302-303. doi: 10.1038/s41409-021-01529-x. Epub 2021 Nov 23. No abstract available. PMID 34815518

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from 2 transplant centers willing to participate signed an Institutional Review Board approved Informed Consent Form and had eligibility for enrollment evaluated. If a participant's eligibility was confirmed they were enrolled into the study. The first participant was enrolled in December 2019, and the last participant was enrolled in January 2020.
Period: Overall Study
Arm/Group | T-Guard Treatment
Started | 3
Initiated T-Guard Treatment | 3
Completed | 0
Not Completed | 3
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: years] | 36.0 [31.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR)
Description: Complete Response at Day 28 is defined as a score of 0 for the GVHD staging in all evaluable organs at the Day 28 visit along with freedom from additional systemic therapy for treatment of acute GVHD.
Time Frame: Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 3
Participants | 0

2. Secondary Outcome: Duration of Complete Response (DoCR)
Description: Evaluate the duration of complete response (DoCR) Early Trial Closure.
Time Frame: Through Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival (OS)
Description: Estimate the overall survival (OS) at Day 30.
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 3
Participants | 3

4. Secondary Outcome: Overall Response Rate (CR or Partial Response (PR))
Description: Estimate the overall response rate (CR or partial response (PR)) at Days 14, 28, and 56.
Time Frame: Days 14, 28, and 56
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

5. Secondary Outcome: Proportions of CR, PR, Mixed Response (MR), no Response (NR) and Progression
Description: Describe proportions of CR, PR, mixed response (MR), no response (NR), and progression of aGVHD at Days 7, 14, 28, and 56.
Time Frame: Days 7, 14, 28, and 56
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Non-Relapse Mortality (NRM)
Description: Estimate the cumulative incidence of non-relapse mortality (NRM) at Days 100 and 180.
Time Frame: Days 100 and 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Relapse-free Survival
Description: Estimate relapse-free survival at Day 180.
Time Frame: Days 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

8. Secondary Outcome: GVHD-free Survival
Description: Estimate GVHD-free survival at Days 90 and 180
Time Frame: Days 90 and 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

9. Secondary Outcome: Cumulative Incidence of Chronic GVHD
Description: Estimate the cumulative incidence of chronic GVHD (cGVHD) at Day 180
Time Frame: Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

10. Secondary Outcome: Cumulative Incidence of Disease Relapse/Progression
Description: Estimate the cumulative incidence of disease relapse/progression at Day 180
Time Frame: Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

11. Secondary Outcome: Incidence of Systemic Infections
Description: Describe the incidence of systemic infections
Time Frame: initiation of T-Guard to 28 days post-last dose
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

12. Secondary Outcome: Incidence of Toxicities
Description: Describe the incidence of CTCAE v5 Grade 3-5 toxicities
Time Frame: initiation of T-Guard to 28 days post-last dose
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

13. Secondary Outcome: Pharmacokinetics of T-Guard - Cinf
Description: Observed and model-predicted concentration of T-Guard at the end of infusion
Time Frame: Before each infusion & at the following post-infusion timepoints: 4, 5, 6, 8 & 24 hours for the 1st infusion; 4, 6 & 24 hours for the 2nd & 3rd infusions; 4, 6, 24 & 48 hours for the 4th infusion (infusions occur within the time frame of Day 0 to Day 14)
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

14. Secondary Outcome: Pharmacokinetics of T-Guard - CL
Description: Systemic clearance of T-Guard
Time Frame: as for outcome 13
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

15. Secondary Outcome: Pharmacokinetics of T-Guard - AUC
Description: Model-predicted area under the curve from the start of the current infusion until the next infusion or until 48 hours following for the last infusion
Time Frame: as for outcome 13
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

16. Secondary Outcome: Pharmacokinetics of T-Guard - t1/2
Description: Model-predicted terminal half-life of T-Guard
Time Frame: as for outcome 13
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

17. Secondary Outcome: Pharmacokinetics of T-Guard - Vc
Description: Volume of the central compartment
Time Frame: as for outcome 13
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

18. Secondary Outcome: Immunogenicity
Description: Assess the immunogenicity of T-Guard via ADA responses in the form of human anti-SPV-T3a-RTA and anti-WT1-RTA -antibodies evaluated in serum samples
Time Frame: Baseline, Days 7, 14, 28, 90, and 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

19. Other Pre Specified Outcome: Corticosteroid Dose
Description: Corticosteroid-dose (measured in prednisone-equivalent) at baseline, Days 28 and 56 post initiation of T- Guard therapy.
Time Frame: Baseline, Days 28 and 56
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

20. Other Pre Specified Outcome: Rate of Near-CR
Description: Estimate the rate of near-CR (i.e. CR in GI and Liver with only Stage 1 Skin) at Days 28 and 56 post initiation of T- Guard therapy
Time Frame: Days 28 and 56
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

21. Other Pre Specified Outcome: Discontinuation of Systemic Steroids
Description: Describe discontinuation of systemic steroids by Day 180 post initiation of T-Guard therapy
Time Frame: Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

22. Other Pre Specified Outcome: Incidence of CMV Reactivation
Description: Estimate the incidence of CMV reactivation requiring therapy by Day 180 post initiation of T-Guard Therapy
Time Frame: Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

23. Other Pre Specified Outcome: Incidence of EBV-associated Lymphoproliferative Disorder or EBV Reactivation
Description: Estimate the incidence of Epstein-Barr Virus (EBV)- associate lymphoproliferative disorder or EBV reactivation requiring therapy with rituximab by Day 180 post initiation of T-Guard therapy
Time Frame: Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

24. Other Pre Specified Outcome: Incidence of IMP-related SAEs
Description: Describe the incidence of Investigational Medicinal Product (IMP) related SAEs
Time Frame: Through Day 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

25. Other Pre Specified Outcome: T-cell Subsets and NK Cells
Description: The evolution of specific cell populations over the 180 day follow-up period and, in particular, T-Guard's effect in depleting targeted T cell and NK cell subsets as well as its impact on relevant non-target populations (B cells, monocytes and dendritic cells), will be evaluated.
Time Frame: Baseline and Days 0, 2, 4, 6, 14, 28, 56, 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

26. Other Pre Specified Outcome: Acute GVHD Biomarkers
Description: Serum ST2 and Regenerating Family Member 3 Alpha (REG3α) concentrations and urine 3- Indoxyl Sulfate (3-IS) concentrations will be used to estimate the probability of NRM at Day 180 post-assessment for each patient. The proportion of patients with high risk biomarker status (defined as estimated NRM greater than 0.29) will be described at each time point.
Time Frame: Baseline and Days 7, 14, 28
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

27. Other Pre Specified Outcome: Patient-reported Outcomes Using a Subset of the PROMIS Measures
Description: Describe changes in patient-reported outcomes (PROs) using a subset of the PROMIS measures from baseline to Days 28, 56, and 180 post initiation of T- Guard therapy
Time Frame: Baseline and Days 28, 56, 180
Population: Study stopped as safety stopping guideline was met.
Arm/Group | T-Guard Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: The study has recruited only 3 SR-aGVHD patients who were treated with T-Guard therapy (2 received the full four doses and 1 received only three doses) during a short period of 69 days.
Description: The adverse event collection followed the clinicaltrials.gov definitions.
Arm/Group | T-Guard Treatment
All-Cause Mortality (participants affected / at risk) | 3/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Guard Treatment (N=3)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) — Grade 3
Cardiac arrest after septic shock (Cardiac disorders) | 1 (1) — Grade 4
Aspergillus pulmonary infection (Infections and infestations) | 3 (4) — Grade 4
Sepsis (Infections and infestations) | 1 (1) — Grade 5
Metapneumovirus infection (Infections and infestations) | 1 (1) — Grade 5
Staphylococcal sepsis (Infections and infestations) | 1 (1) — Grade 5
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Acute kidney injury (Renal and urinary disorders) | 1 (1) — Grade 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T-Guard Treatment (N=3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Differential white blood cell count abnormal (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Septic Shock (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to the early trial closure and limited study population, only a subset of the protocol-specified planned analyses were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agree to the disclosure requirements in a Protocol Rider. This states that the BMT CTN DCC will lead on the initial study Publication, and for any subsequent study Publication, with either a) the advance review of Sponsor or b) two years after the completion of the Study at all Study Sites, the DCC, Participating Sites, and Principal Investigators may publicly disclose or submit for Publication an article, poster or other material that includes analysis of the study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/19/NCT04128319/Prot_SAP_000.pdf